CLINICAL TRIAL: NCT05075564
Title: An Open-Label, Multicenter, First-in-Human, Dose-Escalation, Phase 1 Study of ES002023 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ES002023 (Anti-CD39 Antibody) in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES002023-1001
Record Dates: First submitted 2021-09-21; First posted 2021-10-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 dose escalation (Experimental): ES002023 doses will be escalated in patients with advanced solid tumors with approximately 30 subjects.
  Interventions: Drug: Part 1 ES002023
- Part 2 dose expansion (Experimental): Part 2 of the study will consist of 3 expansion cohorts for pancreatic ductal adenocarcinoma (Cohort 2A), NSCLC (Cohort 2B), and colorectal adenocarcinoma (Cohort 2C) with 10 subjects per expansion cohort respectively at the recommended optimal biological dose determined in Part 1 dose escalation.
  Interventions: Drug: Part 2 ES002023

INTERVENTIONS:
Drug: Part 1 ES002023 — ES002023 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Part 1 dose escalation
Drug: Part 2 ES002023 — ES002023 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Part 2 dose expansion

SUMMARY:
The purpose of this first-in-human, open-label, multicenter, non-randomized study is to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary clinical activity of ES002023 in patients with advanced solid tumors that are relapsed or refractory to standard therapies.

DETAILED DESCRIPTION:
ES002023 is a recombinant humanized IgG1 monoclonal antibody (mAb) that specifically targets the human ectonucleoside triphosphate diphosphohydrolase-1 (ENTPD1, CD39, UniprotKB: P49961). ES002023 is generated using classic hybridoma technology with an attenuated effector domain (Fc) based on human IgG1. ES002023 binding to CD39 inhibits the enzyme activity of ectonucleoside triphosphate diphosphohydrolase, which can result in the stabilization of pro-inflammatory extracellular ATP (eATP) and the restoration of antitumor immunity by impairing the accumulation of immune suppressive adenosine within the tumor microenvironment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Part 1: Histological or cytological documentation of unresectable locally advanced or metastatic solid tumors, if 1) disease has progressed despite standard therapy, and no further standard therapy exists; or 2) standard therapy has proven to be ineffective, intolerable, or is considered inappropriate.

   Part 2: Histological or cytological documentation of pancreatic ductal adenocarcinoma (Cohort 2A), NSCLC (Cohort 2B), or colorectal adenocarcinoma (Cohort 2C), with unresectable locally advanced or metastatic disease, if 1) disease has progressed despite standard therapy, and no further standard therapy exists; or 2) standard therapy has proven to be ineffective, intolerable, or is considered inappropriate.
3. Provide tumor tissue samples obtained from the initial diagnosis to study entry.
4. At least one measurable lesion per RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.
6. Life expectancy of at least 12 weeks.
7. Adequate hematologic, hepatic and renal functions
8. Male and female subjects of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception

Key Exclusion Criteria:

1. Any prior therapy targeting CD39, CD73, or adenosine A2A receptor.
2. Receipt of any investigational agents or devices within 4 weeks prior to the first dose of study drug.
3. Prior treatment with the following therapies:

   * Anticancer therapy within 30 days or 5 half-lives of the drug prior to the first dose of study drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered. Exception: hormonal and/or hormonal replacement therapy.
   * A wash out of at least 2 weeks before the start of study drug for radiation to the extremities and 4 weeks for radiation to the chest, brain, or visceral organs is required.
4. Prior allogeneic or autologous bone marrow transplantation or solid organ transplantation.
5. Toxicity from previous anticancer treatment
6. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug.
7. Subjects who received transfusion of blood products (including platelets or red blood cells), G-CSF, GM-CSF, recombinant erythropoietin, or recombinant thrombopoietin within 14 days prior to the first dose of study treatment.
8. Major surgery within 4 weeks prior to the first dose of study treatment.
9. Live vaccine therapies within 4 weeks prior to the first dose of study treatment.
10. Recent history of allergen desensitization therapy within 4 weeks prior to the first dose of study treatment.
11. Allergy or sensitivity to ES002023 or known allergies to CHO-produced antibodies
12. Invasive malignancy or history of invasive malignancy other than disease under study within the last two years
13. CNS metastases
14. Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications
15. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
16. Active infection requiring systemic therapy, known human immunodeficiency virus (HIV) infection, or positive test for hepatitis B active infection (HBsAg) or hepatitis C active infection (hepatitis C antibody).
17. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
18. History or evidence of cardiac abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
The frequency and severity of adverse events of ES002023 | 1-3 years
  Adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
The Maximum Tolerated Dose (MTD), Optimal Biological Dose (OBD) and/or the Recommended Phase 2 Dose (RP2D) of ES002023 | 1-3 years
  The MTD, OBD and/or RP2D of ES002023 will be determined

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of ES002023 | 1-3 years
  Maximum observed serum concentration (Cmax) of ES002023 will be measured.
Trough observed serum concentration (Ctrough) of ES002023 | 1-3 years
  Trough observed serum concentration (Ctrough)of ES002023 will be measured.
Area under the serum concentration time curve (AUC) of ES002023 | 1-3 years
  Area under the serum concentration time curve (AUC) of ES002023 will be measured.
Time to Cmax (Tmax) of ES002023 | 1-3 years
  Time to Cmax (Tmax) of ES002023 will be measured.
The terminal elimination half life of ES002023 | 1-3 years
  The terminal elimination half-life (t 1/2) of ES002023 will be measured.
The clearance of ES002023 | 1-3 years
  A pharmacokinetic measurement of the volume of plasma from which ES002023 is completely removed per unit time.
The volume of distribution of ES002023 | 1-3 years
  The amount of of ES002023 in the body divided by the plasma concentration will be measured.
The immunogenicity of ES002023 | 1-3 years
  The presence and the frequency of anti-drug antibodies (ADA) against ES002023 will be measured.
The antitumor activity of ES002023 | 1-3 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Elpiscience Biopharma, Ltd.
Locations (7):
- United States (7):
  - HonorHealth, Scottsdale, Arizona
  - Fayetteville Oncology, Fayetteville, Arkansas
  - UCLA, Los Angeles, California
  - Sarah Cannon Research Institute, Orlando, Florida
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NEXT Austin, Austin, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No